CLINICAL TRIAL: NCT05254548
Title: A Single-center, Open-label, Four-period, Fixed-sequence Study to Investigate the Effect of Single and Repeated Oral Doses of ACT-539313 on the Pharmacokinetics of Flurbiprofen, Omeprazole, Midazolam, and Their Respective Metabolites in Healthy Subjects
Brief Title: A Study to Investigate the Effect of Single and Repeated Oral Doses of ACT-539313 on What the Body Does to Flurbiprofen, Omeprazole, Midazolam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ID-082-103; 2021-006214-36 (EudraCT Number)
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Healthy
MeSH Terms: interventions — ACT-539313; Flurbiprofen; Omeprazole; Midazolam

STUDY DESIGN:
Intervention Model Description: Four-period, fixed-sequence drug-drug interaction study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT-539313 with or without a standard combination (probe substrate) (Experimental): Treatment arm has 4 in-house treatment periods. In Treatment Period 1, participants will receive a single oral dose of the standardized combination (probe substrate: containing flurbiprofen [50 mg], midazolam [2 mg] and omeprazole 20 [mg]) on Day 1. Participants will be discharged from the study site on Day 2 and will be re-admitted on Day 7. In Treatment Period 2 (morning of Day 8) a first oral dose of 100 mg ACT-539313 will be administered. One hour later a single oral dose of the probe substrate will be administered. In the evening of Day 8, a second oral dose of 100 mg ACT-539313 will be administered. During Treatment Period 3 (morning of Day 9, ending on the evening of Day 14) oral doses of 100 mg ACT-539313 will be administered in the morning and evening. In Treatment Period 4 (Day 15), a single oral dose of 100 mg ACT-539313 together with the probe substrate will be administered. The participants will receive the last dose of ACT-539313 in the evening of Day 15.
  Interventions: Drug: ACT-539313; Drug: Flurbiprofen; Drug: Omeprazole; Drug: Midazolam

INTERVENTIONS:
Drug: ACT-539313 — 100 mg ACT-539313 (hard capsules) will be administered twice per day in period 2 (morning and evening of Day 8), period 3 (morning and evening of Day 9 to 14) and period 4 (morning and evening of Day 15).
Drug: Flurbiprofen — One daily dose of flurbiprofen 50 mg will be administered in period 1 (morning of Day 1), period 2 (morning of Day 8), and period 4 (morning of Day 15).
Drug: Omeprazole — A single dose of omeprazole 20 mg will be administered in period 1 (morning of Day 1), period 2 (morning of Day 8), and period 4 (morning of Day 15).
Drug: Midazolam — A single dose of midazolam 2 mg will be administered in period 1 (morning of Day 1), period 2 (morning of Day 8), and period 4 (morning of Day 15).

SUMMARY:
A study to investigate the effect of single and repeated oral doses of ACT-539313 on what the body does to flurbiprofen, omeprazole, midazolam in healthy participants.

DETAILED DESCRIPTION:
A screening evaluation will be performed within 3 to 28 days (or within 10 to 28 days for women of childbearing potential) before first study treatment administration. Prior to any screening assessment, participants must sign the informed consent form.

Eligibility will be based on the results of the Screening and Day -1 assessments.

The participants will be confined to the study site from the morning of Day -1 until the morning of Day 2, from the morning of Day 7 until the morning of Day 9 and from the morning of Day 14 until the morning of Day 16. Participants will return to the study site for the End of Study examination on Day 17.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the participant prior to any study-mandated procedure.
* Healthy male or female subjects aged between 18 and 45 years (inclusive) at Screening.
* Body Mass Index of 18.5 to 28.0 kg/m2 (inclusive) at Screening.
* Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1. They must consistently and correctly use (from Screening, during the entire study, and for at least 30 days after study treatment intake) a highly effective method of contraception with a failure rate of < 1% per year, be sexually inactive, or have a vasectomized partner. If a hormonal contraceptive is used, it must have been initiated at least 1 month before treatment administration.
* Women of non-childbearing potential, i.e., postmenopausal (defined as 12 consecutive months with no menses without an alternative medical cause, confirmed by a FSH test), with previous bilateral salpingectomy, bilateral salpingo-oophorectomy or hysterectomy, or with premature ovarian failure (confirmed by a specialist), XY genotype, Turner syndrome, uterine agenesis.
* 12-lead ECG (including QT: < 450 milliseconds [for males] and < 470 milliseconds [for females] without clinically relevant abnormalities, measured after 5 min in the supine position at Screening and on Day -1.

Exclusion Criteria:

* Pregnant or lactating women.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry, and urinalysis, i.e. outside the reference ranges (< 0.9 lower limit of normal and > 1.1 upper limit of normal; except for relevant hepatic parameters [Alanine Aminotransferase (ALT), Aspartate Aminotransferase Test (AST), bilirubin] which must not exceed the upper limit of normal), at Screening and on Day -1.
* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment(s) (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Acute, ongoing, recurrent, or chronic systemic disease with the ability to interfere with the evaluation of the study results.
* Prior history of severe respiratory failure, acute respiratory depression, or sleep apnea.
* Prior history of peptic ulcer disease and/or gastrointestinal bleeding.
* Prior history of asthma, urticaria, or other allergic type reactions after taking acetylsalicylic acid or other NSAIDs.
* History of cardiovascular thrombotic events (including myocardial infarction and stroke) and coronary artery bypass graft surgery.
* Participation in a clinical study involving study treatment administered within 3 months (or 5 t 1/2 of the study treatment administered [whichever is longer]) prior to screening or in more than 4 clinical studies within 1 year prior to Screening.
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St. John's Wort, homeopathic preparations, vitamins, and minerals; with the exception of ibuprofen [1200 mg/day] or paracetamol [up to 1500 mg/day] up until Day -1) within 3 weeks (or 5 t1/2 [whichever is longer]) prior to first study treatment administration.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of each probe substrate: flurbiprofen, midazolam and omeprazole. | Pre-dose through to 24 hours post-dose.
  In periods 1, 2 and 4 the plasma pharmacokinetic parameters of flurbiprofen, omeprazole, and midazolam will be derived by non-compartmental analysis of the plasma concentration-time profiles. Plasma pharmacokinetic samples will be collected at multiple predefined time points to analyze probe substrate: flurbiprofen, midazolam and omeprazole concentrations.
Time to reach Cmax (tmax) of each probe substrate: flurbiprofen, midazolam and omeprazole. | Pre-dose through to 24 hours post-dose.
  In periods 1, 2 and 4 the plasma pharmacokinetic parameters of flurbiprofen, omeprazole, and midazolam will be derived by non-compartmental analysis of the plasma concentration-time profiles. Plasma pharmacokinetic samples will be collected at multiple predefined time points to analyze probe substrate: flurbiprofen, midazolam and omeprazole concentrations.
The area under the plasma concentration-time curve from zero to 24 hours (AUC0-24) of flurbiprofen, midazolam and omeprazole. | Pre-dose through to 24 hours post-dose.
  In periods 1, 2 and 4 the plasma pharmacokinetic parameters of flurbiprofen, omeprazole, and midazolam will be derived by non-compartmental analysis of the plasma concentration-time profiles. Plasma pharmacokinetic samples will be collected at multiple predefined time points to analyze probe substrate: flurbiprofen, midazolam and omeprazole concentrations.
The terminal elimination half-life (t½) of each probe substrate: flurbiprofen, midazolam and omeprazole. | Pre-dose through to 24 hours post-dose.
  In periods 1, 2 and 4 the plasma pharmacokinetic parameters of flurbiprofen, omeprazole, and midazolam will be derived by non-compartmental analysis of the plasma concentration-time profiles. Plasma pharmacokinetic samples will be collected at multiple predefined time points to analyze probe substrate: flurbiprofen, midazolam and omeprazole concentrations.
ACT-539313 trough plasma concentrations (Ctrough) | Pre-dose through to 10 days after first dose.
  In periods 2, 3 and 4 the plasma pharmacokinetic parameters of ACT-539313 will be measured prior to the next dose being administered in the morning.

OTHER OUTCOMES:
Treatment-emergent adverse events | From study treatment administration on Day 1 up to last assessment at End of Study (Day 17).
  All adverse events will be collected, however, adverse events occurring during the in-between period (from end of period 1 up to first study treatment administration in period 2, are not considered as treatment-emergent adverse events.
Maximum plasma concentration (Cmax) of ACT-539313 | Pre-dose through to 24 hours post-dose.
  In periods 2 (Day 8 and 9) and period 4 (Day 15, 16 and 17) the plasma pharmacokinetic parameters of ACT-539313 will be derived by non-compartmental analysis of the plasma concentration-time profiles. Cmax will be analyzed in periods 2 and 4 with the administration of probe substrate. In period 4 the Cmax will be determined after steady state ACT-539313 concentrations have been reached.
Time to reach Cmax (tmax) of ACT-539313 | Pre-dose through to 24 hours after first dose.
  In periods 2 (Day 8 and 9) and period 4 (Day 15, 16 and 17) the plasma pharmacokinetic parameters of ACT-539313 will be derived by non-compartmental analysis of the plasma concentration-time profiles. tmax will be analyzed in periods 2 and 4 with the administration of probe substrate. In period 4 the tmax will be determined after steady state ACT-539313 concentrations have been reached.
Area under the plasma concentration-time curve [AUC(tau)] of ACT-539313 | Pre-dose through to 240 hours after first dose.
  In periods 2 (Day 8 and 9), period 3 (Day 10 to Day 15) and period 4 (Day 15, 16 and 17) plasma pharmacokinetic samples will be collected at multiple predefined time points to analyze ACT-539313 concentrations. AUC(tau) will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berger B, Kaufmann P, Berse M, Treiber A, Grignaschi N, Dingemanse J. Effect of nivasorexant (ACT-539313), a selective orexin-1-receptor antagonist, on multiple cytochrome P450 probe substrates in vitro and in vivo using a cocktail approach in healthy subjects. Pharmacol Res Perspect. 2023 Oct;11(5):e01143. doi: 10.1002/prp2.1143. PMID 37800597